CLINICAL TRIAL: NCT02610543
Title: A Randomized, Double-blind, Placebo-controlled, Proof-of-concept Study to Evaluate the Efficacy of UCB5857 Over 12 Weeks in Subjects With Primary Sjögren's Syndrome
Brief Title: UCB Proof of Concept Study in Patients With Primary Sjögren's Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study stopped prematurely due to enrolment challenges.
Sponsor: UCB Celltech (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SS0004; 2014-004523-51 (EudraCT Number)
Record Dates: First submitted 2015-11-18; First posted 2015-11-20 (Estimated); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Primary Sjögren's Syndrome
Keywords: Primary Sjögren's Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- UCB5857 (Experimental): UCB5857 once daily for 12 weeks
  Interventions: Drug: UCB5857
- Placebo (Placebo Comparator): Placebo once daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: UCB5857 — Active Substance: UCB5857 Pharmaceutical form: Capsule Concentration: 5 mg, 10 mg, 30 mg Route of administration: oral
  Arms: UCB5857
Drug: Placebo — Active substance: Placebo Pharmaceutical Form: Capsule Route of administration: oral
  Arms: Placebo

SUMMARY:
This is a Phase 2, multicenter, double-blind, placebo-controlled, 12-week proof-of-concept study to assess the efficacy, safety, and tolerability of UCB5857 in subjects with primary Sjögren's Syndrome (pSS).

The primary objective of this study is to evaluate the efficacy on overall disease activity and safety of UCB5857 added to current treatment relative to placebo in subjects with pSS.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be between 18 years and 75 years of age
* Women of childbearing potential must agree to use a highly effective method of birth control during the study and for a period of 3 months after their final dose of study drug. Women not agreeing to use birth control must be of non-childbearing potential defined as; permanently sterile, congenitally sterile or postmenopausal for at least 2 years prior to Screening (Visit 1). Women of childbearing potential are required to have a serum pregnancy test taken at Screening (Visit 1), which is confirmed to be negative by urine testing prior to the first dose of study drug at Week 1 (Visit 2) Male subjects with a partner of childbearing potential must be willing to use a condom when sexually active during the study and for 3 months after the last dose of study drug In addition female partner of childbearing potential of male subject must be willing to use a highly effective method of contraception for duration of study and for 3 months after last dose of study drug
* Subject must meet the 2002 AECG (American-European Consensus Group) criteria for Primary Sjӧgren's Syndrome
* Subject must have a serum test positive for anti-SSA/Ro (Ro-52 or Ro-60) and/or anti SSB/La autoantibodies

Exclusion Criteria:

* Subject has a diagnosis of any other autoimmune disease, ie, secondary Sjögren's syndrome (eg, rheumatoid arthritis, systemic lupus erythematosus
* Subject has a diagnosis of any other sicca syndrome (eg, history of head and neck radiation treatment, sarcoidosis chronic graft-versus-host disease)
* Subject has significant fibromyalgia syndrome as defined by the American College of Rheumatology 2010 classification criteria
* Subject has significant depression as defined by the 5th edition of the Diagnostic and Statistical Manual of Mental Disorders
* Subject has oral candidiasis
* Subject is female and is breast-feeding, pregnant, or plans to become pregnant or to start breastfeeding during the study or within 3 months after the final dose of the investigational medicinal product (IMP)
* Subject has evidence of an immunosuppressive state, including human immunodeficiency virus (HIV) infection, hypogammaglobulinemias, T-cell deficiencies, or human T-cell leukemia virus type 1 (HTLV-1)

  o Positive testing for HIV-1/2 at Screening (Visit 1)
* Subject has a history of chronic infections, including but not limited to concurrent acute or chronic viral hepatitis B (HBV) or hepatitis C (HCV)

  * Positive testing for HBV at Screening (Visit 1)
  * Positive testing for HCV at Screening (Visit 1)
* A subject with a history of a recent serious or life-threatening infection or any current signs or symptoms that may indicate a significant infection at Screening (Visit 1) to randomization, as per the Investigator's clinical judgment is also excluded Subject must have completed any prior anti-infective therapy prior to the first dose of study drug with the exception of anti-infectives taken specifically for the treatment of acne, rosacea, onychomycosis, or vaginal yeast infections; for the prophylaxis of urinary tract infections; or prophylaxis for pre-surgical or pre-procedural reasons (including dental procedures). Note: minocycline may not be used for these purposes
* Subject is at a particularly high risk of significant infection due to their lifestyle and/or occupation
* Subject has received intranasal influenza vaccine within the 8 weeks prior to Screening (Visit 1)
* Subject has significant hematologic abnormalities of hemoglobin <10.0 g/dL, or white blood cell (WBC) <2000 /mm^3, or absolute neutrophil count <1000 /mm^3, or platelets <100,000 /mm^3 at Screening (Visit 1)
* Subject has a history of cancer

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-09-07 (Actual); Study Completion 2017-12-05 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to Week 12 in the European League Against Rheumatism Sjögren's Syndrome Disease Activity Index (ESSDAI) | Week 12
  The ESSDAI is a physician administered questionnaire containing 12 organ-specific domains designed to measure disease activity

SECONDARY OUTCOMES:
Change from Baseline to Week 4 in the European League Against Rheumatism Sjögren's Syndrome Disease Activity Index (ESSDAI) | Week 4
  The ESSDAI is a physician administered questionnaire containing 12 organ-specific domains designed to measure disease activity
Change from Baseline to Week 8 in the European League Against Rheumatism Sjögren's Syndrome Disease Activity Index (ESSDAI) | Week 8
  The ESSDAI is a physician administered questionnaire containing 12 organ-specific domains designed to measure disease activity
Change from Baseline to Week 4 in the EULAR Sjögren's Syndrome Patient Response Index (ESSPRI) | Week 4
  The ESSPRI is a patient completed questionnaire to assess subjective patient symptoms, which includes 3 domains (dryness, limb pain and fatigue)
Change from Baseline to Week 8 in the EULAR Sjögren's Syndrome Patient Response Index (ESSPRI) | Week 8
  The ESSPRI is a patient completed questionnaire to assess subjective patient symptoms, which includes 3 domains (dryness, limb pain and fatigue)
Change from Baseline to Week 12 in the EULAR Sjögren's Syndrome Patient Response Index (ESSPRI) | Week 12
  The ESSPRI is a patient completed questionnaire to assess subjective patient symptoms, which includes 3 domains (dryness, limb pain and fatigue)
Change from Baseline to Week 4 in the stimulated salivary flow | Week 4
  The stimulated salivary flow test evaluates the status of salivary glands and the production of saliva. Saliva is collected into a graduated container after gustatory provocation with a stimulant
Change from Baseline to Week 8 in the stimulated salivary flow | Week 8
  The stimulated salivary flow test evaluates the status of salivary glands and the production of saliva. Saliva is collected into a graduated container after gustatory provocation with a stimulant
Change from Baseline to Week 12 in the stimulated salivary flow | Week 12
  The stimulated salivary flow test evaluates the status of salivary glands and the production of saliva. Saliva is collected into a graduated container after gustatory provocation with a stimulant
Change from Baseline to Week 4 in the unstimulated salivary flow | Week 4
  The unstimulated salivary flow test evaluates the status of salivary glands and the production of saliva. Saliva is collected into a graduated container without gustatory provocation
Change from Baseline to Week 8 in the unstimulated salivary flow | Week 8
  The unstimulated salivary flow test evaluates the status of salivary glands and the production of saliva. Saliva is collected into a graduated container without gustatory provocation.
Change from Baseline to Week 12 in the unstimulated salivary flow | Week 12
  The unstimulated salivary flow test evaluates the status of salivary glands and the production of saliva. Saliva is collected into a graduated container without gustatory provocation
Change in sum total tear secretion from Baseline to Week 12 measured by Schirmer´s I test(without anesthesia) | Week 12
  The Schirmer's test measures basic tear function. A 35 mm x 5mm size paper strip is inserted into each eye for a period of 5 minutes to measure the production of tears.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — +18445992273 (UCB)
Locations (14):
- France (3):
  - Ss0004 34, Brest
  - Ss0004 30, Le Kremlin-Bicêtre
  - Ss0004 35, Strasbourg
- Italy (3):
  - Ss0004 20, L’Aquila
  - Ss0004 21, Palermo
  - Ss0004 22, Udine
- Spain (2):
  - Ss0004 42, Córdoba
  - Ss0004 40, Villajoyosa
- Ss0004 50, Stockholm, Sweden
- United Kingdom (5):
  - Ss0004 01, Birmingham
  - Ss0004 05, Essex
  - Ss0004 04, Leeds
  - Ss0004 03, Newcastle upon Tyne
  - Ss0004 02, Swindon

REFERENCES:
- [Result] Juarez M, Diaz N, Johnston GI, Nayar S, Payne A, Helmer E, Cain D, Williams P, Devauchelle-Pensec V, Fisher BA, Giacomelli R, Gottenberg JE, Guggino G, Kvarnstrom M, Mariette X, Ng WF, Rosas J, Sanchez Burson J, Triolo G, Barone F, Bowman SJ. A phase 2 randomized, double-blind, placebo-controlled, proof-of-concept study of oral seletalisib in primary Sjogren's syndrome. Rheumatology (Oxford). 2021 Mar 2;60(3):1364-1375. doi: 10.1093/rheumatology/keaa410. PMID 32949140